CLINICAL TRIAL: NCT02588443
Title: Phase I Study of Neo-adjuvant RO7009789 Alone or Neo-adjuvant RO7009789 Plus Nab-Paclitaxel and Gemcitabine Followed by Adjuvant RO7009789 Plus Nab-Paclitaxel and Gemcitabine for Patients With Newly Diagnosed Resectable Pancreatic Carcinoma
Brief Title: Study of Neo-adjuvant RO7009789 Alone or Neo-adjuvant RO7009789 Plus Nab-Paclitaxel and Gemcitabine Followed by Adjuvant RO7009789 Plus Nab-Paclitaxel and Gemcitabine for Patients With Newly Diagnosed Resectable Pancreatic Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: UPCC 20214
Record Dates: First submitted 2015-10-21; First posted 2015-10-27 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1 (Experimental): Arm I provides one dose of RO70097890 as a single agent in the neoadjuvant setting. Patients will recover from any toxicities and will then have their disease surgically resected. After recovery from surgery patients will proceed to adjuvant therapy which will include nab-paclitaxel 125mg/m2 and gemcitabine 1000mg/m2 on days 1,8 and 15 of a 28 day cycle along with RO7009789 0.2mg/kg on day 3 of each cycle. Four cycles of adjuvant therapy will be given. All medications are administered intravenously.
  Interventions: Drug: RO70097890; Drug: nab-paclitaxel; Drug: gemcitabine
- Arm2 (Experimental): Arm II provides one dose of RO7009789 two days after one dose of nab-paclitaxel and one dose of gemcitabine prior to surgery. Nab-paclitaxel and gemcitabine are given on day 1. RO7009789 will be given on day 3. Patients will recover from any toxicities and will then have their disease surgically resected. Patients will receive four cycles of these same medications in an adjuvant fashion after recovering from surgical resection. A cycle will consist of nab-paclitaxel (125mg/m²), gemcitabine (1000mg/m²) given on days 1,8 and 15 of a 28 day cycle along with RO7009789 0.2mg/kg on day 3 of each cycle.
  Interventions: Drug: RO70097890; Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: RO70097890
Drug: nab-paclitaxel
Drug: gemcitabine

SUMMARY:
The main purpose of this study is to learn if adding the investigational drug RO7009789 (anti-CD40) to nab-paclitaxel and gemcitabine both before surgery and after surgery is safe, feasible, and beneficial to patients with pancreatic cancer. This study also intends to look at blood and tissue samples to help doctors better understand the role of the immune system in fighting cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of primary adenocarcinoma of the pancreas
* Surgically eligible for tumor resection with curative intent
* Age ≥18 years
* ECOG PS 0 or 1
* Adequate bone marrow function (ANC ≥1,500; Hgb >9; Plt >100)
* Adequate renal function (Cr <1.5 ULN)
* Total bilirubin ≤1.5 x ULN; and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN (values post biliary stenting allowed for eligibility).
* Signed, written informed consent

Exclusion Criteria:

* Non ductal adenocarcinomas, neuroendocrine neoplasms, cystic tumors of the pancreas such as cystadenomas, cystadenocarcinomas and solid pseudopapillary neoplasms. In addition, adenocarcinomas arising from duodenum, distal bile duct, and ampulla will also be excluded.
* Patients with M1 disease or a history of M1 disease.
* Patients with any type of recurrent pancreatic adenocarcinoma
* Prior therapy such as chemotherapy or radiation therapy or anti-tumor experimental therapy for pancreatic cancer
* Previous treatment with any other compound that targets CD40
* Concurrent treatment with any anticancer agent outside of this protocol
* Prior allogeneic bone marrow transplant
* History of autoimmune disorder, including type 1 diabetes mellitus, pemphigus vulgaris, systemic mastocytosis, systemic lupus erythromatosis, dermatomyositis/polymyositis, rheumatoid arthritis, systemic sclerosis, Sjörgen's syndrome, vasculitis/arteritis, Behcet's syndrome, autoimmune thyroiditis, multiple sclerosis, or uveitis,. (Vitiligo is allowed)
* History (within the previous year) of stroke or transient ischemic attack, unstable angina, myocardial infarction, congestive heart failure
* History of deep venous thrombosis or migratory thrombophlebitis (Trousseau);
* Hereditary or acquired coagulopathies (e.g., hemophilia, von Willebrand disease, or cancer-associated DIC)
* Prior allergic reactions attributed to other monoclonal antibodies
* Concurrent or planned concurrent treatment with systemic high dose (immunosuppressive) corticosteroids or treatment with systemic corticosteroids within 4 weeks of baseline
* Treatment on another therapeutic clinical trial within 4 weeks of enrollment in this trial
* Concurrent or planned concurrent treatment with anticoagulants such as Coumadin or heparin, except to maintain patency of in-dwelling catheters
* Ongoing or active infection; treatment with systemic antibiotics or antifungals for ongoing or recurrent infection (topical use of antibiotics or antifungals is allowed)
* Pregnancy or breast-feeding - female patients must be surgically sterile, be post-menopausal, or must agree to use effective contraception during the period of therapy and for 90 days following the last dose of RO7009789. All female patients with reproductive potential must have a negative pregnancy test prior to enrollment. Women or men of reproductive potential may not participate unless they agree to use an effective contraceptive method. Female patients should not become pregnant while participating in this research study or for 90 days following therapy. Male patients should not father a child while in this research study or for 90 days following therapy.
* Other uncontrolled, concurrent illness that would preclude study participation; or, psychiatric illness or social challenges that would entail unreasonable risk or preclude informed consent or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vonderheide, MD, DPhil, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States